CLINICAL TRIAL: NCT04515966
Title: Randomized Controlled Trial of Ultrasound-guided Steroid Injection Versus Wrist Splint in Patients With Carpal Tunnel Syndrome
Brief Title: A Comparison of Ultrasound-guided Steroid Injection With Wrist Splint in Carpal Tunnel Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mercy Health Ohio (Other)
Responsible Party: Principal Investigator, Roy Morcos, Professor, Family and Community Medicine, Mercy Health Ohio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-006
Record Dates: First submitted 2020-08-05; First posted 2020-08-17 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: wrist splint; steroid injection; median nerve ultrasound
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Lidocaine; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound-guided steroid injection (Active Comparator): Participants with CTS who meet the inclusion criteria are randomized to two groups. One group (or arm) will receive an ultrasound-guided steroid injection in the vicinity of the median nerve within the carpal tunnel. A total 1 ml of injectate consisting of 0.5 ml of depo-Medrol (methylprednisolone acetate 40mg/ml) and 0.5 mL of 1% lidocaine is injected into the carpal tunnel under ultrasound guidance to deliver it into the target area. After completion of the injection, the distal carpal tunnel is scanned to ensure injectate distribution within the distal aspect of the carpal tunnel.
  Interventions: Drug: Methylprednisolone Injection [Solu-Medrol]
- Wrist splint (Active Comparator): Participants in this arm are treated with a wrist splint.
  Interventions: Device: wrist splint

INTERVENTIONS:
Drug: Methylprednisolone Injection [Solu-Medrol] — A total 1 ml of injectate consisting of 0.5 ml of depo-Medrol (methylprednisolone acetate 40mg/ml) and 0.5 mL of 1% lidocaine will be injected into the carpal tunnel under ultrasound guidance to deliver it into the target area. After completion of the injection, the distal carpal tunnel is scanned to ensure injectate distribution within the distal aspect of the carpal tunnel.
  Other Names: Lidocaine, 1% solution
  Arms: Ultrasound-guided steroid injection
Device: wrist splint — A standard wrist splint
  Arms: Wrist splint

SUMMARY:
Carpal Tunnel Syndrome (CTS) is caused by compression of a nerve called the median nerve as it travels through a narrow tunnel within the wrist on its way to the hand. Compression of the median nerve causes numbness, tingling, pain and weakness of the hand and fingers. CTS is usually treated with rest or a change in the activity level. It can also be treated with a splint that limits bending of the hand and wrist. Other treatments include a steroid injection near the median nerve. Surgery can be performed if the symptoms are severe or persistent.

Compression of the median nerve can cause swelling that may be observed with ultrasound of the wrist. Ultrasound can also be used to help guide the needle to inject the steroid solution in close proximity to the median nerve while avoiding injury to the nerve.

The investigators plan to compare the effectiveness of a splint and an ultrasound-guided steroid injection in the treatment of mild to moderate CTS. Individuals with CTS who agree to participate, will be randomly assigned to two groups. One group will be treated with a splint and the other with a steroid injection performed under ultrasound guidance. The severity of CTS symptoms will be determined prior to beginning the study and also at 6 weeks, 3 months, 6 months and 1 year following each of the two treatment interventions. The median nerve size (diameter) will be measured in all participants prior to beginning the study and also following both treatment interventions at 6 weeks, 3 months, 6 months and 1 year.

At the conclusion of the study, the investigators will determine which of the two treatments, splint or steroid injection, is more effective in alleviating CTS symptoms. The investigators will also determine if either or both treatments result in a change in swelling of the median nerve as measured by ultrasound.

DETAILED DESCRIPTION:
The purpose of the study is to determine which of two commonly used therapeutic interventions for the treatment of carpal tunnel syndrome (CTS), steroid injection or wrist splint, is more effective in alleviating symptoms. The protocol has been approved by the Medical Research Committee and by the Institutional Review Board, Mercy Health, Youngstown.

The steroid injection will be administered under ultrasound guidance to ensure proper placement of the needle in close proximity to the median nerve within the carpal tunnel and to minimize the risk of direct trauma to the nerve.

Candidates for the study will be individuals with CTS presenting to primary care offices located in the Boardman, Ohio area. Following a detailed explanation of the study purpose and protocol, those individuals who agree to participate will be asked to sign an informed consent form.

A complete history and physical examination will be performed on all participants to confirm the diagnosis. Additionally, baseline ultrasound measurement of the median nerve cross-sectional area within the carpal tunnel will be performed on all participants. The diagnosis of CTS will be made on clinical grounds, and the CTS-6 evaluation tool will also be used in the diagnostic evaluation. A score above 12 will be considered consistent with CTS. Participants with moderately severe CTS will undergo a nerve conduction study to confirm the diagnosis and exclude early signs of denervation which may require surgical decompression.

Participants will be randomized into two groups of thirty-five patients each; those in group A will undergo ultrasound-guided steroid injection and those in group B will be asked to wear a standard carpal tunnel splint. Participants will be randomly assigned to either intervention group with the use of a computer-generated random sequence of numbers from 1 to 70. The primary investigator (Roy Morcos) will be responsible for maintaining confidential records in a secure location.

The injections will be performed by Dr. Morcos and Dr. Dhungana. Dr. Morcos received training in ultrasonography during a fellowship program and has published on the subject. He has been performing ultrasound examinations and injections for the past 35 years. Dr. Dhungana is an orthopedic surgeon with expertise in carpal tunnel steroid injections.

With the participant seated and the forearm supinated, the wrist is slightly dorsiflexed. The median nerve is identified with real-time ultrasonography and its cross-sectional area measured. Injection near the median nerve within the carpal tunnel is performed under aseptic technique and ultrasound guidance, using a 25-gauge needle to minimize discomfort.

Group A: A mixture of 0.5 ml of depo-Medrol (methylprednisolone acetate 40mg/ml) and 0.5 mL of 1% lidocaine will be injected into the carpal tunnel under ultrasound guidance in close proximity to the median nerve. After completion of the injection, the distal carpal tunnel is scanned to ensure even injectate distribution within the distal aspect of the carpal tunnel.

Group B: Patients in this group will be advised to wear a standard carpal tunnel splint with the hand in neutral position. The splint will be provided to all participants. They will be advised to wear it during the night and most of the time during day.

The median nerve cross-sectional area is measured in all patients at baseline, 6 weeks and 3 months following interventions.

Follow-up is scheduled 6 weeks, 3 months, 6 months and one year. At each follow-up visit, clinical evaluation is obtained using the BCTQ score, which determines the degree of symptomatic severity and functional recovery. A visual analog scale (VAS) for pain, 0 for no pain and 10 for severe unbearable pain, will also be obtained. Follow-up will continue for a year including history and physical examination.

Descriptive statistics will be used to characterize the data using the mean, standard deviation, and median. For parameter with subset scales and values, box and whisker plots will be used to show patterns of parameter behavior. Where levels of measures are appropriate, independent samples t-tests are performed to compare outcomes of each intervention. Where appropriate, a non-parametric test such as the Mann-Whitney U test, is used to assess differences of parameter values both over periods of follow up and between two treatments.

The measures of effect are as follows: Pain, Symptom severity, Functional disability, Median nerve diameter, Median nerve cross sectional area. Three of the parameters are from arbitrary scales consisting of standard questionnaires. Two of the parameters are composite values derived from scores with differing weightings. Two anatomic measures are based on metric measurements obtained by ultrasound. All measures will be taken before treatment and at 6 weeks, 12 weeks, 6 months and 1 year. Based on an assumed BCTS Pain Score treatment effect of 1.5 with standard deviation of 3.0 with 2-sided α of 0.05 and a power of 0.87, the minimum required sample size in each study group is 32. Considering loss to follow-up over a period of one year, the investigators plan to recruit 70 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with typical symptoms of CTS, including nocturnal, postural, or usage-associated paresthesia of the hand
* symptoms persisting for at least 3 months before the study
* Patients with mild to moderate symptoms
* no history of steroid injections in the past
* no history of CT release surgery
* and age 18 to 75.

Exclusion Criteria:

* Thenar atrophy or muscle weakness
* severe CTS
* pregnancy
* hypothyroidism
* diabetes mellitus
* chronic renal failure
* rheumatoid arthritis
* orthopedic or neurological disorders that could mimic CTS such as cervical radiculopathy, polyneuropathy, proximal median nerve entrapment, or thoracic outlet syndrome
* history of distal radius fracture
* anticoagulation
* chronic use of systemic corticosteroids
* known allergy to corticosteroids and local anesthetics.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Carpal tunnel syndrome, Change in symptom severity from baseline to 6 weeks | Baseline, 6 weeks
  Boston Carpal Tunnel Questionnaire (BCTQ) Symptom Severity Scale (SSS). 11 questions with score ranging from 1 (Normal) to 5 (Very Serious). Composite score range 11-55. The score mapping is as follows: 11: Asymptomatic; 12 to 22: Mild; 23 to 33: Moderate; 34 to 44: Severe; 45-55: Very Severe.
  Questionnaire is administered by an investigator.
Carpal tunnel syndrome, Change in functional status from baseline to 6 weeks | Baseline, 6 weeks
  Boston Carpal Tunnel Questionnaire (BCTQ) Functional Status Scale (FSS). 8 questions with score ranging from 1 (No Difficulty) to 5 (Unable to Perform). Composite score range 8-40. The score mapping is as follows: 8: Asymptomatic; 9 to 16: Mild; 17 to 24: Moderate; 25 to 32: Severe; 33-40: Very Severe.
  Questionnaire is administered by an investigator.
Carpal tunnel syndrome, Change in pain assessment from baseline to 6 weeks | Baseline, 6 weeks
  Visual Analog Scale (VAS). A visual pain scale measures a patient's pain intensity. Scale ranging from 0 (No Pain) to 10 (Unbearable Pain) characterized by depictions of facial expressions. The score mapping is as follows: 0: No Pain; 1 to 3: Mild Pain; 4 to 6: Moderate Pain; 7 to 10: Severe Pain
  Assessment is performed by an investigator.

SECONDARY OUTCOMES:
Change in Median Nerve Dimensions | Baseline, 6 weeks, 12 weeks, 6 months, 1 year
  The median nerve dimensions at the carpal tunnel inlet is measured by high-resolution ultrasound. The diameter is measured in millimeters, and cross-sectional area calculated in square millimeters
Carpal tunnel syndrome, Change in symptom severity at 12 weeks, 6 months, 1 year | 12 weeks, 6 months, 1 year
  Boston Carpal Tunnel Questionnaire (BCTQ) Symptom Severity Scale (SSS). 11 questions with score ranging from 1 (Normal) to 5 (Very Serious). Composite score range 11-55. The score mapping is as follows: 11: Asymptomatic; 12 to 22: Mild; 23 to 33: Moderate; 34 to 44: Severe; 45-55: Very Severe.
  Questionnaire is administered by an investigator.
Carpal tunnel syndrome, Change in functional status at 12 weeks, 6 months, 1 year | 12 weeks, 6 months, 1 year
  Boston Carpal Tunnel Questionnaire (BCTQ) Functional Status Scale (FSS). 8 questions with score ranging from 1 (No Difficulty) to 5 (Unable to Perform). Composite score range 8-40. The score mapping is as follows: 8: Asymptomatic; 9 to 16: Mild; 17 to 24: Moderate; 25 to 32: Severe; 33-40: Very Severe.
  Questionnaire is administered by an investigator.
Carpal tunnel syndrome, Change in pain perception at 12 weeks, 6 months, 1 year | 12 weeks, 6 months, 1 year
  Visual Analog Scale (VAS). A visual pain scale measures a patient's pain intensity. Scale ranging from 0 (No Pain) to 10 (Unbearable Pain) characterized by depictions of facial expressions. The score mapping is as follows: 0: No Pain; 1 to 3: Mild Pain; 4 to 6: Moderate Pain; 7 to 10: Severe Pain
  Assessment is performed by an investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Roy N. Morcos, M.D., Principal Investigator — Bon Secours Mercy Health
Locations (1):
- St. Elizabeth Boardman Family Medicine, Boardman, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klauser AS, Halpern EJ, Faschingbauer R, Guerra F, Martinoli C, Gabl MF, Arora R, Bauer T, Sojer M, Loscher WN, Jaschke WR. Bifid median nerve in carpal tunnel syndrome: assessment with US cross-sectional area measurement. Radiology. 2011 Jun;259(3):808-15. doi: 10.1148/radiol.11101644. Epub 2011 Mar 8. PMID 21386049
- [Background] Demircay E, Civelek E, Cansever T, Kabatas S, Yilmaz C. Anatomic variations of the median nerve in the carpal tunnel: a brief review of the literature. Turk Neurosurg. 2011;21(3):388-96. doi: 10.5137/1019-5149.JTN.3073-10.1. PMID 21845577
- [Background] Karadas O, Tok F, Akarsu S, Tekin L, Balaban B. Triamcinolone acetonide vs procaine hydrochloride injection in the management of carpal tunnel syndrome: randomized placebo-controlled study. J Rehabil Med. 2012 Jun;44(7):601-4. doi: 10.2340/16501977-0990. PMID 22674243
- [Background] Tagliafico A, Bodner G, Rosenberg I, Palmieri F, Garello I, Altafini L, Martinoli C. Peripheral nerves: ultrasound-guided interventional procedures. Semin Musculoskelet Radiol. 2010 Nov;14(5):559-66. doi: 10.1055/s-0030-1268066. Epub 2010 Nov 11. PMID 21072732
- [Background] Chesterton LS, Blagojevic-Bucknall M, Burton C, Dziedzic KS, Davenport G, Jowett SM, Myers HL, Oppong R, Rathod-Mistry T, van der Windt DA, Hay EM, Roddy E. The clinical and cost-effectiveness of corticosteroid injection versus night splints for carpal tunnel syndrome (INSTINCTS trial): an open-label, parallel group, randomised controlled trial. Lancet. 2018 Oct 20;392(10156):1423-1433. doi: 10.1016/S0140-6736(18)31572-1. PMID 30343858
- [Background] Padua L, Coraci D, Erra C, Pazzaglia C, Paolasso I, Loreti C, Caliandro P, Hobson-Webb LD. Carpal tunnel syndrome: clinical features, diagnosis, and management. Lancet Neurol. 2016 Nov;15(12):1273-1284. doi: 10.1016/S1474-4422(16)30231-9. Epub 2016 Oct 11. PMID 27751557
- [Background] Middleton SD, Anakwe RE. Carpal tunnel syndrome. BMJ. 2014 Nov 6;349:g6437. doi: 10.1136/bmj.g6437. No abstract available. PMID 25378457
- [Background] Calandruccio JH, Thompson NB. Carpal Tunnel Syndrome: Making Evidence-Based Treatment Decisions. Orthop Clin North Am. 2018 Apr;49(2):223-229. doi: 10.1016/j.ocl.2017.11.009. Epub 2018 Feb 1. PMID 29499823
- [Background] Kim PT, Lee HJ, Kim TG, Jeon IH. Current approaches for carpal tunnel syndrome. Clin Orthop Surg. 2014 Sep;6(3):253-7. doi: 10.4055/cios.2014.6.3.253. Epub 2014 Aug 5. PMID 25177448
- [Background] Jarvik JG, Comstock BA, Kliot M, Turner JA, Chan L, Heagerty PJ, Hollingworth W, Kerrigan CL, Deyo RA. Surgery versus non-surgical therapy for carpal tunnel syndrome: a randomised parallel-group trial. Lancet. 2009 Sep 26;374(9695):1074-81. doi: 10.1016/S0140-6736(09)61517-8. PMID 19782873
- [Background] So H, Chung VCH, Cheng JCK, Yip RML. Local steroid injection versus wrist splinting for carpal tunnel syndrome: A randomized clinical trial. Int J Rheum Dis. 2018 Jan;21(1):102-107. doi: 10.1111/1756-185X.13162. Epub 2017 Sep 13. PMID 28901660
- [Background] Evers S, Bryan AJ, Sanders TL, Selles RW, Gelfman R, Amadio PC. Effectiveness of Ultrasound-Guided Compared to Blind Steroid Injections in the Treatment of Carpal Tunnel Syndrome. Arthritis Care Res (Hoboken). 2017 Jul;69(7):1060-1065. doi: 10.1002/acr.23108. Epub 2017 Jun 8. PMID 27696773
- [Background] Khosrawi S, Emadi M, Mahmoodian AE. Effectiveness of splinting and splinting plus local steroid injection in severe carpal tunnel syndrome: A Randomized control clinical trial. Adv Biomed Res. 2016 Feb 8;5:16. doi: 10.4103/2277-9175.175902. eCollection 2016. PMID 26962518